CLINICAL TRIAL: NCT06379997
Title: Efficacy of Oral Hyaluronic Acid and Collagen Supplementation Compared With Hyaluronic Acid Infiltration Treatment in Rotator Cuff Tendinopathies: A Prospective Study
Brief Title: Oral Supplementation Compared With Hyaluronic Acid Infiltration in Rotator Cuff Tendinopathies
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: I.R.C.C.S. Fondazione Santa Lucia (Other)
Responsible Party: Principal Investigator, Stefano Brunelli, Principal Investigator, MD, I.R.C.C.S. Fondazione Santa Lucia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SANTA LUCIA IRCCS
Record Dates: First submitted 2024-04-18; First posted 2024-04-23 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Tendinitis of Shoulder; Hyaluronic Acid; Dietary Supplements; Shoulder Pain
MeSH Terms: conditions — Shoulder Pain | interventions — Collagen; Hyaluronic Acid; Ascorbic Acid; Manganese

STUDY DESIGN:
Intervention Model Description: The enrolled patients will be randomized in two groups: treated with oral supplements (Group 1 - G1) or with intra-articular hyaluronic acid (Group 2 - G2)
Who Masked: Investigator
Masking Description: Both study groups will undergo assessment using pain and functional scales by a clinician who is blinded to the treatment group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral supplemention (Active Comparator): Assumption of 1 vial/day starting from the day after enrollment for 56 days. This supplement contains Collagen, Hyaluronic Acid, Vitamin C, and Manganese.
  Interventions: Dietary Supplement: Collagen, Hyaluronic Acid, Vitamin C, and Manganese
- Intra-articolar infiltration (Active Comparator): Intra-articular injections of a viscous solution of sodium salt hyaluronic acid (500-730 kDa) in pre-filled 20 mg/2 ml syringes, 1/week for 3 weeks.
  Interventions: Drug: Intra-articular infiltration

INTERVENTIONS:
Dietary Supplement: Collagen, Hyaluronic Acid, Vitamin C, and Manganese — The Group 1 (G1) will begin taking a dietary supplement the day after enrollment.
  Other Names: Tendogenial
  Arms: Oral supplemention
Drug: Intra-articular infiltration — Group 2 (G2) will receive three intra-articular injections once per week for 3 weeks, without ultrasound guidance. The route of administration will be intra-articular via the posterior access route.
  Other Names: Hyalotend
  Arms: Intra-articolar infiltration

SUMMARY:
The present study aims to investigate the effectiveness of oral supplementation with a nutraceutical containing Collagen, Hyaluronic Acid, Vitamin C, and Manganese in functional outcome and pain reduction in cases of shoulder rotator cuff tendinopathy compared to a cycle of intra-articular hyaluronic acid injections.

The project involves the recruitment of 50 adult individuals presenting with shoulder pain and instrumental evidence of rotator cuff tendinopathy. All participants will receive one intra-articular injection of 1 ml of triamcinolone acetonide 40 mg. After the injection, participants will be divided into two groups according to Good Clinical Practice guidelines. One group will begin taking one vial per day for 56 days of an oral supplement containing Hyaluronic Acid, Collagen, Vitamin C, and Manganese (HA-COL) (Tendogenial®, B2Pharma) starting from the day following enrollment (Group 1). The other group will undergo a cycle of 3 intra-articular injections with hyaluronic acid (HA) (Hyalotend®, Fidia) (Group 2).

The hypothesis is that oral supplementation with HA-COL may have the same efficacy as intra-articular hyaluronic acid treatment in reducing pain and improving shoulder functionality.

Functional assessments will be conducted by a clinician unaware of the participants' group assignment. The following assessment scales will be used:

Numeric Rating Scale (NRS) for pain (from 0 to 10), evaluating 3 aspects of pain: 1) pain at rest, 2) nocturnal pain, 3) pain during movement.

Shoulder Disability Questionnaire (SDQ) for functionality.

Assessments will be conducted at the following time points:

T0) Before the administration of corticosteroid intra-articular injection (baseline).

T1) Seven days after the start of HA-COL intake for Group 1 and before the first intra-articular HA injection for Group 2 (T1, seven days from T0).

T2) At mid-cycle of oral HA-COL supplementation for Group 1 (28 days of intake) and seven days after the last HA injection for Group 2 (T2, 21 days from T1).

T3) Follow-up at 28 days from T2, at the end of the 56-day oral treatment cycle for Group 1, and 28 days after the last injection for Group 2 (T3, 56 days from T0).

DETAILED DESCRIPTION:
Background Shoulder pain is a prevalent symptom primarily affecting the adult population, with an incidence of approximately 19 per 1000 and a prevalence ranging from 7 to 26%, particularly affecting women. The primary cause of shoulder pain is rotator cuff pathology, characterized by nocturnal pain and weakness, especially during external rotation and elevation movements of the shoulder, attributable to excessive loading on the cuff tissues. These symptoms often result in disability and functional impairment.

The etiology of rotator cuff pathology appears multifactorial, often associated with chronic age-related degeneration characterized by a reduced ability to synthesize collagen, increased levels of free radicals, and heightened catabolic activity (5). Tendinopathies exhibit widespread structural changes, including increased apoptosis of tenocytes, collagen fiber disintegration leading to a decrease in collagen type I, an increase in collagen type III resulting in a reversal of the collagen I/III ratio, and ineffective neoangiogenesis.

As tendinopathy primarily represents a degenerative condition where the inflammatory component plays a minor role, current therapeutic strategies mainly focus on regenerative approaches. While intra-articular cortisone therapy has historically been utilized to alleviate pain from rotator cuff injuries, its potential detrimental effect on tendon collagen limits its long-term efficacy, rendering cortisone therapy beneficial only in the short term.

Conversely, intra-articular treatment with hyaluronic acid (HA) for rotator cuff injuries appears promising in reducing pain and improving shoulder function. A recent review analyzed 11 studies encompassing a total of 1102 patients. Low to medium molecular weight hyaluronic acids were utilized in these studies, with infiltration performed either via anatomical landmarks or ultrasound guidance, targeting either intra-articular or subacromial sites. Moreover, rare minor side effects (such as pain at the injection site or slight vagal effects) were reported, with no instances of allergic reactions.

Hyaluronic acid (HA) is a carbohydrate, specifically a mucopolysaccharide, naturally present in all living organisms. When unbound to other molecules, it binds to water, imparting a rigid viscous 'jelly-like' quality. HA serves as an integral component of synovial fluid, crucial for joint chondroprotection, and constitutes a significant portion of the tendon extracellular matrix.

Upon injection into a joint, HA diminishes cytokine-induced responses and reduces synovial inflammation, ultimately relieving pain and enhancing joint function. Notably, preclinical in vitro and in vivo studies have demonstrated that exogenous peritendinous HA possesses the ability to inhibit fibroblast activity and diminish the proinflammatory M1 activation state of macrophages.

Observations of improved lubrication, chondroprotection, and enhanced synovial fluid characteristics have also been reported. Additionally, HA facilitates tenocyte regeneration, modulates the ratio of collagen type I/III, and mitigates apoptosis and impaired angiogenesis.

It is important to note that in most studies, HA was not injected directly into the degenerated tendon but rather near and/or into the joint space. While it can be speculated that alterations in synovial fluid may positively impact the tendon itself, it remains plausible that clinical improvement could be secondary to the favorable effects on concomitant arthrosis frequently associated with the condition.

Rationale for Dietary Supplementation of Collagen and HA:

Tendons primarily comprise cells, predominantly tenoblasts along with endothelial cells and some chondrocytes, as well as proteoglycans, notably decorin and hyaluronic acid, and collagen, primarily type I. The tendon exhibits a highly organized extracellular matrix wherein collagen molecules assemble into filamentous collagen fibrils (formed by microfibrils), which further aggregate to constitute collagen fibers, the principal structural components.

Various reviews have assessed the effectiveness of oral collagen supplementation in enhancing tendon structure. Particularly, a review highlights that some studies have demonstrated promising clinical implications of collagen peptide supplementation in the prevention and treatment of tendinopathies, although conclusive evidence is still lacking. Another review indicates that collagen supplementation alongside physical training significantly influences pain relief, increased cross-sectional area, and tendon thickness . From a joint perspective, collagen supplementation enhances mobility and functionality while reducing pain.

Oral supplementation of hyaluronic acid has predominantly been investigated for its effects on joints. For instance, it has been found effective in ameliorating pain and enhancing the quality of life in patients with knee arthrosis, with sustained effects observed at 2 months . Furthermore, the combined administration of HA and collagen orally has shown to improve functional recovery in patients following anterior cruciate ligament reconstruction, with evidence from resonance imaging indicating improved neoligament maturation.

Experimental design In order to conduct this study, we will recruit 50 patients with rotator cuff injuries from the outpatient clinic of the Santa Lucia Foundation. A physiatrist from the clinic, participating in the project, will explain the study to the enrolled individuals and obtain their informed consent.

The enrolled patients will undergo infiltrative treatment with corticosteroids (Triamcinolone acetonide 40 mg, 1 vial - Kenacort®, BRISTOL-MYERS SQUIBB S.r.l.).

The enrolled patients will be randomized in 2 groups: oral supplements (Group 1 - G1) or intra-articular hyaluronic acid (Group 2 - G2).

The Experimental Group (G1) will begin taking a supplement called Tendogenial® (B2Pharma S.r.l.) the day after enrollment. This supplement contains Collagen, Hyaluronic Acid, Vitamin C, and Manganese. Each day for 28 days, participants in G1 will consume one vial of Tendogenial®.

Group 2 (G2) will receive three intra-articular injections of Hyalotend® (Fidia), a viscous solution of sodium salt hyaluronic acid (500-730 kDa) obtained by bacterial fermentation in buffered saline. The injections will be administered without ultrasound guidance, using pre-filled 20 mg/2 ml syringes. The route of administration will be intra-articular via the posterior access route.

Participants will be advised to take only paracetamol as needed for pain relief. Additionally, they will be instructed not to undergo physiotherapy during the study period. Any participants who undergo physiotherapy or receive other analgesic therapies during the study will be excluded from the statistical analysis.

Inclusion Criteria:

Persistent shoulder pain lasting for at least 2 months, unresponsive to conservative treatment (nonsteroidal anti-inflammatory drugs [NSAIDs] and rehabilitation).

Ultrasound or MRI evidence of a rotator cuff lesion without complete tendon rupture.

Limited active range of motion (ROM) in the shoulder. Age between 30 and 80 years. Willingness to provide informed consent to participate in the study.

Exclusion Criteria:

Traumatic shoulder injury as the cause of pain. History of shoulder dislocation, fracture, or previous shoulder surgery. Presence of signs indicating ligamentous instability. Severe shoulder arthrosis, adhesive capsulitis, or calcific tendinitis. Previous infiltrative treatment with corticosteroids, hyaluronic acid, or collagen within the past 6 months.

Diagnosis of rheumatic or neoplastic diseases. Ongoing therapy with anticoagulants. Cervical radiculopathy. Pregnancy. History of heart, kidney, or liver failure. Cognitive impairment.

Both study groups will undergo assessment using pain and functional scales by a clinician who is blinded to the treatment group.

In addition to providing informed consent to participate in the study, participants will also sign a consent form specifically for infiltration, prepared by the Santa Lucia Foundation. Any adverse reactions or side effects experienced by participants will be documented and reported.

ELIGIBILITY:
Inclusion Criteria:

* Persistent shoulder pain lasting for at least 2 months unresponsive to conservative treatment (nonsteroidal anti-inflammatory drugs [NSAIDs] and rehabilitation)
* Ultrasound or MRI evidence of a rotator cuff lesion without complete tendon rupture
* Limited active range of motion (ROM) in the shoulder

Exclusion Criteria:

* Traumatic shoulder injury as the cause of pain
* History of shoulder dislocation, fracture, or previous shoulder surgery
* Presence of signs indicating ligamentous instability
* Severe shoulder arthrosis, adhesive capsulitis, or calcific tendinitis
* Previous infiltrative treatment with corticosteroids, hyaluronic acid, or collagen within the past 6 months
* Diagnosis of rheumatic or neoplastic diseases
* Ongoing therapy with anticoagulants
* Cervical radiculopathy
* Pregnancy
* History of heart, kidney, or liver failure
* Cognitive impairment

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-08-10 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Numeric rating scale (NRS) | 1) (T0 - baseline). 2) Before the first administration of intra-articular HA for Group 2 and at seven days from the initiation of HA-COL for Group 1 (T1, seven days from T0). 3) At seven days fo
  Change from baseline NRS at 1 weeks and at 4 weeks and at 8 weeks. NRS is a 10-point scale grading the pain at rest, during movement and during night-time

SECONDARY OUTCOMES:
Shoulder Disability Questionnaire (SDQ) for shoulder functionality | 1) (T0 - baseline). 2) Before the first administration of intra-articular HA for Group 2 and at seven days from the initiation of HA-COL for Group 1 (T1, seven days from T0). 3) At seven days fo
  Change from baseline SDQ at 1 weeks and at 4 weeks and at 8 weeks. The SDQ is a self-assessment scale comprising 22 items designed to gauge functional limitations in daily activities and participation in social engagements among patients with shoulder disorders. Each item requires a YES/NO response, with YES scored as 1. A higher total score (up to 22) indicates greater disability attributed to the shoulder pathology

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Brunelli, MD, Study Director — I.R.C.C.S. Fondazione Santa Lucia, Roma, Italy
Locations (1):
- I.R.C.C.S. Fondazione Santa Lucia, Roma, RM, Italy

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices)
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 5 years following article publication
Access Criteria: Proposals should be directed to the personal corrisponding author's mail address.

REFERENCES:
- [Background] Luime JJ, Koes BW, Hendriksen IJ, Burdorf A, Verhagen AP, Miedema HS, Verhaar JA. Prevalence and incidence of shoulder pain in the general population; a systematic review. Scand J Rheumatol. 2004;33(2):73-81. doi: 10.1080/03009740310004667. PMID 15163107
- [Background] Greving K, Dorrestijn O, Winters JC, Groenhof F, van der Meer K, Stevens M, Diercks RL. Incidence, prevalence, and consultation rates of shoulder complaints in general practice. Scand J Rheumatol. 2012 Mar;41(2):150-5. doi: 10.3109/03009742.2011.605390. Epub 2011 Sep 21. PMID 21936616
- [Background] Dabija DI, Gao C, Edwards TL, Kuhn JE, Jain NB. Genetic and familial predisposition to rotator cuff disease: a systematic review. J Shoulder Elbow Surg. 2017 Jun;26(6):1103-1112. doi: 10.1016/j.jse.2016.11.038. Epub 2017 Feb 2. PMID 28162885
- [Background] Herrmann SJ, Izadpanah K, Sudkamp NP, Strohm PC. Tears of the rotator cuff. Causes--diagnosis--treatment. Acta Chir Orthop Traumatol Cech. 2014;81(4):256-66. PMID 25137495
- [Background] Via AG, De Cupis M, Spoliti M, Oliva F. Clinical and biological aspects of rotator cuff tears. Muscles Ligaments Tendons J. 2013 Jul 9;3(2):70-9. doi: 10.11138/mltj/2013.3.2.070. Print 2013 Apr. PMID 23888289
- [Background] Ackermann PW, Renstrom P. Tendinopathy in sport. Sports Health. 2012 May;4(3):193-201. doi: 10.1177/1941738112440957. PMID 23016086
- [Background] Coombes BK, Bisset L, Vicenzino B. Efficacy and safety of corticosteroid injections and other injections for management of tendinopathy: a systematic review of randomised controlled trials. Lancet. 2010 Nov 20;376(9754):1751-67. doi: 10.1016/S0140-6736(10)61160-9. Epub 2010 Oct 21. PMID 20970844
- [Background] van der Worp H, van den Akker-Scheek I, van Schie H, Zwerver J. ESWT for tendinopathy: technology and clinical implications. Knee Surg Sports Traumatol Arthrosc. 2013 Jun;21(6):1451-8. doi: 10.1007/s00167-012-2009-3. Epub 2012 May 1. PMID 22547246
- [Background] Osti L, Buda M, Buono AD, Osti R, Massari L. Clinical evidence in the treatment of rotator cuff tears with hyaluronic acid. Muscles Ligaments Tendons J. 2016 Feb 13;5(4):270-5. doi: 10.11138/mltj/2015.5.4.270. eCollection 2015 Oct-Dec. PMID 26958534
- [Background] Lee LC, Lieu FK, Lee HL, Tung TH. Effectiveness of hyaluronic acid administration in treating adhesive capsulitis of the shoulder: a systematic review of randomized controlled trials. Biomed Res Int. 2015;2015:314120. doi: 10.1155/2015/314120. Epub 2015 Jan 31. PMID 25802845
- [Background] Salamanna F, Frizziero A, Pagani S, Giavaresi G, Curzi D, Falcieri E, Marini M, Abruzzo PM, Martini L, Fini M. Metabolic and cytoprotective effects of in vivo peri-patellar hyaluronic acid injections in cultured tenocytes. Connect Tissue Res. 2015 Feb;56(1):35-43. doi: 10.3109/03008207.2014.979166. Epub 2014 Nov 13. PMID 25333747
- [Background] Iwata H. Pharmacologic and clinical aspects of intraarticular injection of hyaluronate. Clin Orthop Relat Res. 1993 Apr;(289):285-91. PMID 8472428
- [Background] Oliva F, Marsilio E, Asparago G, Frizziero A, Berardi AC, Maffulli N. The Impact of Hyaluronic Acid on Tendon Physiology and Its Clinical Application in Tendinopathies. Cells. 2021 Nov 9;10(11):3081. doi: 10.3390/cells10113081. PMID 34831304
- [Background] Abate M, Schiavone C, Salini V. The use of hyaluronic acid after tendon surgery and in tendinopathies. Biomed Res Int. 2014;2014:783632. doi: 10.1155/2014/783632. Epub 2014 May 8. PMID 24895610
- [Background] Franchi M, Trire A, Quaranta M, Orsini E, Ottani V. Collagen structure of tendon relates to function. ScientificWorldJournal. 2007 Mar 30;7:404-20. doi: 10.1100/tsw.2007.92. PMID 17450305
- [Background] Hijlkema A, Roozenboom C, Mensink M, Zwerver J. The impact of nutrition on tendon health and tendinopathy: a systematic review. J Int Soc Sports Nutr. 2022 Aug 3;19(1):474-504. doi: 10.1080/15502783.2022.2104130. eCollection 2022. PMID 35937777
- [Background] Boldt KS, Olson BL, Thiele RM. Effects of Collagen and Exercise on Tendon Properties and Pain: A Critically Appraised Topic. J Sport Rehabil. 2023 Sep 27;32(8):938-941. doi: 10.1123/jsr.2023-0115. Print 2023 Nov 1. PMID 37758259
- [Background] Campos LD, Santos Junior VA, Pimentel JD, Carrega GLF, Cazarin CBB. Collagen supplementation in skin and orthopedic diseases: A review of the literature. Heliyon. 2023 Mar 28;9(4):e14961. doi: 10.1016/j.heliyon.2023.e14961. eCollection 2023 Apr. PMID 37064452
- [Background] Kalman DS, Heimer M, Valdeon A, Schwartz H, Sheldon E. Effect of a natural extract of chicken combs with a high content of hyaluronic acid (Hyal-Joint) on pain relief and quality of life in subjects with knee osteoarthritis: a pilot randomized double-blind placebo-controlled trial. Nutr J. 2008 Jan 21;7:3. doi: 10.1186/1475-2891-7-3. PMID 18208600
- [Background] Lopez-Vidriero E, Olive-Vilas R, Lopez-Capape D, Varela-Sende L, Lopez-Vidriero R, Til-Perez L. Efficacy and Tolerability of Progen, a Nutritional Supplement Based on Innovative Plasma Proteins, in ACL Reconstruction: A Multicenter Randomized Controlled Trial. Orthop J Sports Med. 2019 Feb 27;7(2):2325967119827237. doi: 10.1177/2325967119827237. eCollection 2019 Feb. PMID 30834280
- [Background] Leon-Lopez A, Morales-Penaloza A, Martinez-Juarez VM, Vargas-Torres A, Zeugolis DI, Aguirre-Alvarez G. Hydrolyzed Collagen-Sources and Applications. Molecules. 2019 Nov 7;24(22):4031. doi: 10.3390/molecules24224031. PMID 31703345
- [Background] Clark KL, Sebastianelli W, Flechsenhar KR, Aukermann DF, Meza F, Millard RL, Deitch JR, Sherbondy PS, Albert A. 24-Week study on the use of collagen hydrolysate as a dietary supplement in athletes with activity-related joint pain. Curr Med Res Opin. 2008 May;24(5):1485-96. doi: 10.1185/030079908x291967. Epub 2008 Apr 15. PMID 18416885
- [Background] Noriega-Gonzalez DC, Drobnic F, Caballero-Garcia A, Roche E, Perez-Valdecantos D, Cordova A. Effect of Vitamin C on Tendinopathy Recovery: A Scoping Review. Nutrients. 2022 Jun 27;14(13):2663. doi: 10.3390/nu14132663. PMID 35807843
- [Background] Ozgen M, Firat S, Sarsan A, Topuz O, Ardic F, Baydemir C. Short- and long-term results of clinical effectiveness of sodium hyaluronate injection in supraspinatus tendinitis. Rheumatol Int. 2012 Jan;32(1):137-44. doi: 10.1007/s00296-010-1577-0. Epub 2010 Jul 31. PMID 20676646
- [Background] Croft P, Pope D, Zonca M, O'Neill T, Silman A. Measurement of shoulder related disability: results of a validation study. Ann Rheum Dis. 1994 Aug;53(8):525-8. doi: 10.1136/ard.53.8.525. PMID 7944638
- [Background] Brindisino F, Pellicciari L, Lorusso M, Pennella D, Padua R, Di Bari M. Cross-cultural adaptation, reliability, and validity of the Italian version of the Shoulder Disability Questionnaire. Musculoskelet Sci Pract. 2020 Apr;46:102123. doi: 10.1016/j.msksp.2020.102123. Epub 2020 Jan 31. PMID 32217269
- [Background] Chou WY, Ko JY, Wang FS, Huang CC, Wong T, Wang CJ, Chang HE. Effect of sodium hyaluronate treatment on rotator cuff lesions without complete tears: a randomized, double-blind, placebo-controlled study. J Shoulder Elbow Surg. 2010 Jun;19(4):557-63. doi: 10.1016/j.jse.2009.08.006. Epub 2009 Dec 5. PMID 19963403
- [Background] Moghtaderi A, Sajadiyeh S, Khosrawi S, Dehghan F, Bateni V. Effect of subacromial sodium hyaluronate injection on rotator cuff disease: A double-blind placebo-controlled clinical trial. Adv Biomed Res. 2013 Nov 30;2:89. doi: 10.4103/2277-9175.122517. eCollection 2013. PMID 24524035
- [Background] Byun SD, Park DH, Choi WD, Lee ZI. Subacromial Bursa Injection of Hyaluronate with Steroid in Patients with Peri-articular Shoulder Disorders. Ann Rehabil Med. 2011 Oct;35(5):664-72. doi: 10.5535/arm.2011.35.5.664. Epub 2011 Oct 31. PMID 22506189